CLINICAL TRIAL: NCT06868771
Title: Studio Sulla Efficacia Di Una Crema Emolliente Contenente Pre E Postbiotici E Niacinamide 4% Nel Trattamento Della Xerosi Cutanea E Del Prurito in Pazienti Oncologici in Trattamento Con Anti-EGFR
Brief Title: Study on the Effectiveness of an Emollient Cream Containing Pre and Postbiotic and Niacinamide 4% in the Treatment of Skin Xerosis and Itching in Oncological Patients Treated with Anti-EGFR
Acronym: PENSANTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Societa Italiana di Dermatologia Medica, Chirurgica, Estetica e di Malattie Sessualmente Trasmesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SID04
Record Dates: First submitted 2023-07-25; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Xerosis Cutis
MeSH Terms: interventions — Therapeutics; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cases (Other): topical treatment with the pre- and postbiotic and niacinamide 4% study preparation
  Interventions: Other: topical treatment with the pre- and postbiotic study preparation and niacinamide 4% and one with the 10% urea-based preparation.
- control (Other): prepared from 10% urea.
  Interventions: Other: topical treatment with the pre- and postbiotic study preparation and niacinamide 4% and one with the 10% urea-based preparation.

INTERVENTIONS:
Other: topical treatment with the pre- and postbiotic study preparation and niacinamide 4% and one with the 10% urea-based preparation. — Application of the topical preparation in both groups will be performed twice a day for a total duration of 3 months.

SUMMARY:
Study on the Effectiveness of an Emollient Cream Containing Pre and Postbiotic and Niacinamide 4% in the Treatment of Skin Xerosis and Itching in Oncological Patients Treated With Anti-EGFR.

DETAILED DESCRIPTION:
Epidermal growth factor receptor inhibitors (EGFRi) are drugs approved as treatment options in several solid tumors, such as advanced colon, head-neck, breast and lung cancers, because overexpression or mutation of EGFR is implicated in the pathogenesis of these types of cancer. EGFR, in addition to being expressed by neoplastic cells, is also present constitutively on basal keratinocytes, and its inhibition can determine in these cells apoptotic effects, cell growth inhibition, alteration of physiological cell migration and inflammatory processes through the release of pro-inflammatory cytokines, recruitment of leukocytes and the release of pro-apoptotic molecules.

Among the possible adverse skin events (cae), the papulo-pustular rash is the most frequent in the course of therapy with EGFRi (45-90%). In addition to the papulopustulous rash, xerosis and itching are the main dermatological AE associated with EGFRi therapy, with a significant negative impact on the quality of life (qol) of cancer patients.

The reduction of itching and subsequent scratching can therefore be effective in preventing the exacerbation of skin lesions and improving qol in cancer patients, especially in those who experience intense skin xerosis. Emollients containing urea and ceramides have proved useful in skin hydration in case of cutaneous xerosis and in attenuating the associated itching. However, there are few articles in the literature that compare the moisturizing and antipruritic effects of the various basic components of emollients, especially in patients undergoing oncological treatment with EGFRi.

The goals are to examine the effectiveness of an emollient cream containing the prebiotic α-glucan oligosaccharide, the postbiotic Lactobacillus ferment pure (obtained by patented extraction method BPTech) and niacinamide 4%, in the treatment of xerosis, and to test the effectiveness and superiority of this topical preparation in skin hydration and in soothing pruritic symptoms compared to a 10% urea cream commonly used in clinical practice in patients with skin xerosis.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18 who have been receiving anti-EGFR therapy for more than three months,
2. signature of the informed consent.

Exclusion Criteria:

1. Patients diagnosed with Grade II papulopustulous skin reaction according to the Common Terminology Criteria for Adverse Event (CTCAE) scale at the time of enrolment;
2. concomitant use of emollients and/or steroidal creams;
3. personal history of xerotic pathologies (e.g. lichen, ichthyosis) and/or itching of n.d.d.;
4. inability to provide informed consent or inability to complete the procedures required for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Skin hydration | 3 months
  Evaluation of increased skin hydration by comparing specific epidermal parameters in the RCM at different times.
decrease in surface desquamation | 3 months
  assess the decrease in superficial skin desquamation
clinical evaluation the decrease in the size of the skin grooves | 3 months
  evaluate the decrease in the size of the skin grooves in the stratum corneum at different timepoints
decrease in cellular irregularities | 3 months
  assess the decrease in cellular irregularities in the stratum corneum and the stratum spinous and inflammation in the superficial dermis at different time points
clinical evaluation the increase in the degree of brilliance of the intercheratinocyte space | 3 months
  assess the increase in the degree of brilliance of the intercheratinocyte space in the spinous layer the different timepoints;
changes in the arrangement of collagen fibres in the dermis | 3 months
  assess thickening and changes in the arrangement of collagen fibers in the dermis to the different timepoint

SECONDARY OUTCOMES:
skin problems on quality of life (SKINDEX-16) | 3 months
  incidence of skin problems on quality of life
Visual Analogue Scale (VAS) | 3 months
  itch scale

CONTACTS AND LOCATIONS:
Overall Officials: Ketty MD Peris, Principal Investigator — IRCCS FONDAZIONE POLICLINICO GEMELLI
Locations (1):
- Irccs Fondazione Policlinico Gemelli, Roma, ROMA, Italy

IPD SHARING:
Plan to Share IPD: No